CLINICAL TRIAL: NCT04845269
Title: Post-Stroke Osteopathy: Characterization of Fractures and Changes in the Bone Microstructure After Ischemic Stroke or TIA
Brief Title: Post-Stroke Osteopathy
Status: Completed | Type: Observational
Sponsor: VASCage GmbH (Other)
Collaborators: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: VASC-E3-2020-06
Record Dates: First submitted 2021-04-07; First posted 2021-04-14 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Stroke (CVA) or TIA; Fracture; Fall
Keywords: high-resolution peripheral quantitative Computer Tomography; Bone microstructure
MeSH Terms: conditions — Stroke; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CTX1 und CTX 2, Osteocalcin, TRAP5b, Bone Alkaline Phosphatase, Sclerostin, Periostin, RANKL-OPG-Ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The sudden biomechanical inactivation, direct neuro-humoral effects and sustained systemic stress reaction, which commonly occur after stroke or TIA, all may be of relevance in triggering alterations in bone metabolism and remodelling of bone microstructure.

The objectives of this observational pilot study are to characterize falls and fractures and their circumstances (sex and age specific incidence, time course, risk conditions, localization) in ischemic stroke patients, study changes in the bone microstructure after ischemic stroke supported by high-resolution peripheral quantitative Computer Tomography, unravel a molecular mechanisms underlying the increased fracture risk (focus on Wnt-signaling and ß-adrenergic projection), establish risk factors to estimate the risk of falls based on information from gait analysis as well as construct deep learning algorithms to identify bone microstructure parameters for predicting fractures.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion in the STROKE-CARD Registry Study
* Modified Rankin Scale (mRS) < 5
* Provision of signed and dated informed consent form
* Willingness to comply with all study procedures and ability to participate in the study over the complete study duration

Exclusion Criteria:

* Persistent motor deficit before the onset event
* Not able to walk without walking aid or not able to put the full bodyweight on either leg before the onset event
* Medical history of stroke
* Premedication with Corticosteroids for more than 6 Weeks or Pioglitazone or Bisphosphonate within the last 12 months
* Limb amputation
* BMI < 18,5 kg/m2 or > 35 kg/m2
* Present or previous fracture in the distal Radius or Tibia interfering with HR-pQCT
* Movement disorder interfering with HR-pQCT imaging
* Women of childbearing potential

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As a sub-study of the STROKE-CARD Registry Study the source population will be all patients treated at the Department of Neurology Innsbruck (Austria) for stroke and included in the STROKE-CARD Registry Study. The target study population for the Post-Stroke Osteopathy Study will be all patients included in the STROKE-CARD Registry Study (clinicaltrials.gov ID NCT04582825).
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with and without fractures | 12 months

OTHER OUTCOMES:
Changes in imaging bone structure between the baseline and follow-up in all extremities as measured by quantitative CT imaging | 12 months
Number and circumstances (housing situation, concomitant medication, level of immobility,...) of falls between baseline and one-year follow-up | 12 months
  Due to the observational nature of the study, these outcome parameters will be published with descriptive statistics
Change in blood bone biomarkers (as mentioned before) between baseline and follow-up | 12 months
  CTX1 und CTX 2, Osteocalcin, TRAP5b, Bone Alkaline Phosphatase, Sclerostin, Periostin, RANKL-OPG-Ratio
Circumstances (housing situation, concomitant medication, level of immobility,...) of fractures during the twelve-month follow up | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Knoflach, Assoz.Prof. Priv.-Doz. Dr., Principal Investigator — Medical University of Innsbruck, Department of Neurology
Locations (1):
- Medical University of Innsbruck, Department of Neurology, Innsbruck, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] GBD 2017 Causes of Death Collaborators. Global, regional, and national age-sex-specific mortality for 282 causes of death in 195 countries and territories, 1980-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1736-1788. doi: 10.1016/S0140-6736(18)32203-7. Epub 2018 Nov 8. PMID 30496103
- [Background] Yuan ZC, Mo H, Guan J, He JL, Wu ZJ. Risk of hip fracture following stroke, a meta-analysis of 13 cohort studies. Osteoporos Int. 2016 Sep;27(9):2673-2679. doi: 10.1007/s00198-016-3603-x. Epub 2016 Apr 22. PMID 27101998
- [Background] Ramnemark A, Nyberg L, Borssen B, Olsson T, Gustafson Y. Fractures after stroke. Osteoporos Int. 1998;8(1):92-5. doi: 10.1007/s001980050053. PMID 9692083
- [Background] Ramnemark A, Nilsson M, Borssen B, Gustafson Y. Stroke, a major and increasing risk factor for femoral neck fracture. Stroke. 2000 Jul;31(7):1572-7. doi: 10.1161/01.str.31.7.1572. PMID 10884456
- [Background] Ramnemark A, Nyberg L, Lorentzon R, Olsson T, Gustafson Y. Hemiosteoporosis after severe stroke, independent of changes in body composition and weight. Stroke. 1999 Apr;30(4):755-60. doi: 10.1161/01.str.30.4.755. PMID 10187874
- [Background] Carda S, Cisari C, Invernizzi M, Bevilacqua M. Osteoporosis after stroke: a review of the causes and potential treatments. Cerebrovasc Dis. 2009;28(2):191-200. doi: 10.1159/000226578. Epub 2009 Jun 30. PMID 19571530
- [Background] Poole KE, Vedi S, Debiram I, Rose C, Power J, Loveridge N, Warburton EA, Reeve J, Compston J. Bone structure and remodelling in stroke patients: early effects of zoledronate. Bone. 2009 Apr;44(4):629-33. doi: 10.1016/j.bone.2008.11.017. Epub 2008 Dec 11. PMID 19121416
- [Background] Ramnemark A, Nyberg L, Lorentzon R, Englund U, Gustafson Y. Progressive hemiosteoporosis on the paretic side and increased bone mineral density in the nonparetic arm the first year after severe stroke. Osteoporos Int. 1999;9(3):269-75. doi: 10.1007/s001980050147. PMID 10450417
- See also: Datasheet of the µCT — https://www.scanco.ch/images/Brochures/xtremectIIB-v4.pdf